CLINICAL TRIAL: NCT01319396
Title: Performance Validation of a Non-contact Breathing Frequency Monitor (Model BM07)
Status: Completed | Type: Observational
Sponsor: ResMed (Industry)
Responsible Party: Sponsor
Other Study IDs: BM07_8DTS
Record Dates: First submitted 2011-03-16; First posted 2011-03-21 (Estimated); Results first posted 2011-08-15 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Unspecified Threat to Breathing
Keywords: breathing rate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare the accuracy of the BiancaMed BM07 breathing frequency indicator device with the respiration rate measured by a SomnoScreen RC Easy device on 20+ human volunteers. This is being carried out in support of a 510(k) submission.

DETAILED DESCRIPTION:
The purpose of this study is to compare the accuracy of the BiancaMed BM07 breathing frequency indicator device with the respiration rate measured by a SomnoScreen RC Easy device on 20+ human volunteers. This is being carried out in support of a 510(k) submission.

* The BM07 is a non-contact device, using radio frequency (RF) range measurement to detect the chest wall motion, and thus the respiration rate. The BM07 is a CE Class IIa cleared device.
* The SomnoScreen RC Easy is both a CE and FDA (K060708) cleared device, used as an overnight, portable sleep recorder. One of its inputs is a pair of chest respiration effort bands that can be used to record the breathing rate of the subject.
* The human volunteers are selected to be a range of age, body mass index (BMI) and gender so as to cover a broad cross section of the population. BMI, gender and age are features that might affect the performance of the RF reflected signal:

  * High BMI or low BMI could affect the skin RF reflectivity.
  * High BMI may mask chest wall movement during breathing.
  * The thinner skin often associated with increasing age may affect RF reflectivity.
  * Female breast tissue may affect RF reflectivity or mask chest wall movement.

The target performance is an agreement between the BM07 and the Somnoscreen of +/- 5 breaths per minute. This target has been selected based upon a literature review, in particular:

* Lim et al: Respiratory Rate Measurement in Adults - How Reliable is it?
* Droitcour PhD Thesis: Non-Contact Measurement of Heart and Respiration Rates with a Single-Chip Microwave Doppler Radar.

There is no risk to the subjects as the RF energy emitted by the BM07 is much less than that of either a mobile phone bluetooth or a domestic WLAN router.

The testing is to be carried out on volunteer human subjects, who sign a consent form. The locations of testing are Dublin, Ireland and Belfast, UK.

The testing comprises the subjects sitting still for periods of 2 minutes whilst recordings are taken from both the BM07 and Somnoscreen. The test configurations are ranges from the BM07 to subject of 0.5, 1.0 & 1.5m and 1.0m with a thick folded duvet (overblanket/comforter) covering the subject to represent them wearing thick outdoor winter clothing. Each test configuration is carried out twice, making a total of 8 test recordings per subject.

The first 2 volunteers will be used to confirm that the maximum effective range of the BM07 is at least 1.5 m and that the target aspect of the subject (ie the sensor being in front, to one side and from behind) does not affect the ability of the BM07 to detect breathing movement.

This is an Observational study as the subjects are normal healthy volunteers and no intervention can be made as a result of the study measurements

ELIGIBILITY:
Inclusion Criteria:

* volunteer
* consent

Exclusion Criteria: none

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: twenty two plus volunteer subjects, distributed on the follwoing parameters: gender balance: 1/3:2/3 or better. age range: aged 10 years through to senior citizens BMI range: 19 to 40+, or wider
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul D Phillips, MSc, MA, Principal Investigator — ResMed
Locations (1):
- ResMed, Dublin, Ireland

RESULTS

PARTICIPANT FLOW:
Groups:
- 5GHz Sensor Spot Respiration Rate: All participants had the difference in indicated breathing rate measured. The 2 devices were the BM07 5GHz non-contact sensor (device under test) and the Somnoscreen (reference device using chest effort bands)
Period: Overall Study
Arm/Group | 5GHz Sensor Spot Respiration Rate
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- 5.8 GHz Sensor Spot Respiration Rate: All participants had the difference in indicated breathing rate measured. The 2 devices were the BM07 5GHz non-contact sensor (device under test) and the Somnoscreen (reference device using chest effort bands)
Arm/Group | 5.8 GHz Sensor Spot Respiration Rate
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 20
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 16
Region of Enrollment [Number; unit: participants]
  United Kingdom | 9
  Ireland | 15

OUTCOME MEASURES:

1. Primary Outcome: Respiration Rate Accuracy - Mean Difference in Breaths Per Minute Between the BM07 5GHz Sensor and SomnoScreen Devices
Description: The respiration rate measured contemporaneously by the BM07 5GHz sensor and the reference device, SomnoScreen, are compared on a second-by-second basis, over the recording duration. The difference between the two respiration rate measurements (the delta) for all 24 subjects' recordings, in all positions, are plotted on a normal distribution chart, giving 10,542 data points. The distribution chart reveals the mean difference between the two devices' measurements and the Standard Deviation (SD). The measure of success is if the 95% (ie 2SD) of the difference in the respiration rate indicated by the two devices (the delta) is less than 5 breaths per minute. This measure is derived from the peer review paper by Lim et al, cited in the References section
Time Frame: Recording duration of 2 minutes; measurement made after 45 seconds settling time, for at least 60 seconds
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | 5GHz Sensor Spot Respiration Rate
Number analyzed (Participants) | 24
breaths per minute | 0.28 (1.2)

ADVERSE EVENTS:
Time Frame: adverse events were collected during the 2 minute period that participants were taking part in the evaluation
Arm/Group | 5.8 GHz Sensor Spot Respiration Rate
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 0/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5.8 GHz Sensor Spot Respiration Rate (N=24)
General (Respiratory, thoracic and mediastinal disorders) | 0 (0) — The nature of the device is that it is not acting on the subject. It just monitors the general breathing rate whilst the subjects are sitting still. Thus no serious or non serious adverse events were expected and non were reported
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 5.8 GHz Sensor Spot Respiration Rate (N=24)
General (Respiratory, thoracic and mediastinal disorders) | 0 (0) — The nature of the device is that it is not acting on the subject. It just monitors the general breathing rate whilst the subjects are sitting still. No adverse events occurred during the evaluation

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes